CLINICAL TRIAL: NCT00165438
Title: A Prospective Study of Pulmonary Function in Patients With Hodgkin's Disease Receiving Bleomycin-Based Chemotherapy With or Without Mediastinal Irradiation
Brief Title: Pulmonary Function in Patients With Hodgkin's Disease Receiving Bleomycin-Based Chemotherapy
Status: Completed | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Andrea K. Ng, MD, Principal Investigator, Dana-Farber Cancer Institute
Other Study IDs: 01-181
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Hodgkin's Disease
Keywords: Pulmonary function; Bleomycin-based chemotherapy; mediastinal irradiation
MeSH Terms: conditions — Hodgkin Disease | interventions — Respiratory Physiological Phenomena

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Pulmonary Function Tests — Tests include; total lung capacity, vital capacity, functional residual capacity, forced vital capacity, forced expiratory volume in 1 second, carbon monoxide diffusing capacity, pulse oximetry before and after a 6 minute walk and Pulmonary Status and Dyspnea Questionnaire
Procedure: CAT Scan — Obtained at different time points during the study depending upon standard of care chemotherapy treatment

SUMMARY:
The purpose of this study is to find out the impact Bleomycin-containing chemotherapy, given with or without chest radiation therapy, on patients' lung function over time.

DETAILED DESCRIPTION:
* The tests and procedures in this study are part of regular cancer care but this study offers more structured timing of these standard tests.
* Due to the potential lung toxicity associated with bleomycin-based chemotherapy, pulmonary function tests are routinely performed. Pulmonary function tests will be performed by a licensed, registered respiratory therapist and performed prior to the beginning of treatment, between the chemotherapy and radiation therapy (only for patients receiving both chemotherapy and radiation therapy), and at approximately 1 month, 6 months, 1 year and 2 years after the completion of all treatments.
* A CAT scan will be performed prior to the beginning of treatment, and approximately 1 month, 6 months, 1 year and 2 years after the completion of all treatments.
* A self-administered questionnaire will be performed on the days the patient is undergoing pulmonary function tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed classical Hodgkin's disease, with mediastinal involvement
* Bleomycin-based chemotherapy alone or in combination with mediastinal irradiation

Exclusion Criteria:

* Prior chest irradiation
* Mediastinal irradiation received at an outside institution
* Refractory or progressive disease on treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed classic Hodgkin's disease with mediastinal involvement in whom bleomycin-based chemotherapy alone or bleomycin-based chemotherapy and mediastinal irradiation are recommended as initial treatment.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2001-10; Primary Completion 2005-11 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Pulmonary function | 2 years
  Changes in pulmonary function over time

CONTACTS AND LOCATIONS:
Overall Officials: Andrea K. Ng, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts